CLINICAL TRIAL: NCT01184313
Title: Acute Lung Injury After Aortic Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Reija Mikkola/MS, Oulu University
Other Study IDs: Mikkola2010
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-08

CONDITIONS: Lung Injury
Keywords: aortic valve surgery; CPB; lung injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- aortic valve surgery
  Interventions: Procedure: aortic valve surgery with CPB

INTERVENTIONS:
Procedure: aortic valve surgery with CPB — elective aortic valve surgery with CPB

SUMMARY:
The purpose of this prospective, randomized clinical trial is to understand and measure lung injuries caused by CPB in aortic valve surgery.

Study questions:

* Is there any correlation between the release of pro-inflammatory biomarkers and lung injury degree?
* Is there any correlation between oxyhaemodynamic parameters and lung injury degree?
* Is there any correlation between oxyhaemodynamic parameters and the release of pro-inflammatory biomarkers?
* Are budesonide, erdostein and acetylcystein effective in the prevention of lung injuries?

ELIGIBILITY:
Inclusion Criteria:

* elective aortic valve surgery patient
* written consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: elective aortic valve surgery patients in Oulu University hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09

PRIMARY OUTCOMES:
lung injury | within the first 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Reija Mikkola, MS, Principal Investigator — Oulu University Hospital; Fausto Biancari, MD, PhD, Study Director — Oulu University Hospital; Juha Koskenkari, MD, Study Chair — Oulu University Hospital; Vesa Pakanen, MD, Study Chair — Oulu University Hospital; Tatu Juvonen, prof., Study Chair — Oulu University Hospital
Locations (1):
- Oulu University hospital, Oulu, Finland